CLINICAL TRIAL: NCT01623037
Title: Pilot Study of Non-Invasive Fat Layer Reduction in the Flanks of Asian Patients With the CoolCurve+ Applicator
Brief Title: Pilot Study on The Flanks of Asian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA12-006
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2012-06

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CoolSculpting Treatment Group (Experimental): The single arm will include all subjects treated on each flank with the CoolSculpting System and CoolCurve+ applicator. Treatment temperature and duration are defined in the protocol.
  Interventions: Device: The Zeltiq System

INTERVENTIONS:
Device: The Zeltiq System — Non-invasive cooling is applied to the each flank with a defined cooling rate and duration.
  Other Names: Cryolipolysis; Lipolysis

SUMMARY:
This study will evaluate CoolSculpting and the CoolCurve applicator for non-invasive fat reduction in the flanks with sharp body curvature.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the performance of the CoolCurve+ applicator for non-invasive fat layer reduction in flanks for Asian patient population.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects > 18 years of age.
2. Subjects must be of Asian descent.
3. Subject has clearly visible fat on the flanks, which in the investigator's opinion, may benefit from the treatment.
4. Subject has not had weight change exceeding 10 pounds in the preceding month.
5. Subject with body mass index (BMI) up to 25. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
6. Subject with sharp flank curvature that fits well with the CoolCurve+ applicator.
7. Subject agrees to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in their diet or lifestyle during the course of the study.
8. Subject has read and signed a written informed consent form.

Exclusion Criteria

1. Subject has had a surgical procedure(s) in the area of intended treatment.
2. Subject has had an invasive fat reduction procedure (e.g., liposuction, abdominoplasty, mesotherapy) in the area of intended treatment.
3. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 6 months.
4. Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
5. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
6. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
7. Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
8. Subject is taking or has taken diet pills or supplements for weight loss within the past month.
9. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
10. Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
11. Subject is pregnant or intending to become pregnant during the study period (in the next 4 months).
12. Subject is lactating or has been lactating in the past 6 months.
13. Subject is unable or unwilling to comply with the study requirements.
14. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
15. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06-21; Primary Completion 2012-09-21 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Chan, MD, Principal Investigator — Hong Kong Dermatology and Laser Centre
Locations (1):
- Hong Kong Dermatology and Laser Centre, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CoolSculpting Treatment Group: The single arm will include all subjects treated on the each flank with the CoolSculpting System and CoolCurve+ applicator. Treatment temperature and duration are defined in the protocol.
  The Zeltiq System: Non-invasive cooling is applied to the each flank with a defined cooling rate and duration.
Period: Overall Study
Arm/Group | CoolSculpting Treatment Group
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 41.1 [29 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Region of Enrollment [Number; unit: participants]
  Hong Kong | 15
BMI [Mean (Full Range); unit: kg//m^2] | 22.8 [21 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Pre-treatment Images Correctly Identified
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline and pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Success is defined as 70% correct identification of pre-treatment images.
Time Frame: Baseline and 12 weeks post-final treatment
Population: All subjects in the analysis group were treated on each flank with CoolSculpting. Each subject had pre-treatment and post-treatment images taken.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 15
Number analyzed (photos) | 45
photos | 32
Statistical Analysis 1: Comparison: CoolSculpting Treatment Group; Test type: Other; sucess proportion = 71.1, 95% CI 2-sided [55.7 to 83.6]

2. Primary Outcome: Safety of the CoolSculpting and the CoolCurve+ Applicator
Description: The number of device- or procedure-related adverse events will be tabulated for all AEs reported continuously throughout the study, from enrollment to the final 12 week follow-up visit.
Time Frame: Enrollment through 12 weeks post-final treatment
Population: All subjects treated with the CoolSculpting device and CoolCurve+ applicator were included in the population.
Measure: Number; unit: device or procedure-related AE's
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 15
device or procedure-related AE's | 0

3. Secondary Outcome: Subject Satisfaction With the Procedure
Description: Subject satisfaction as assessed by questionnaire administered at 12-weeks post-treatment will be tabulated. The questionnaire will be composed of 5-point Likert scale questions, as well as free-text responses. Subjects will be asked to determine overall satisfaction with the treatment. The choices will be: 1) very unsatisfied; 2) somewhat unsatisfied; 3) neither unsatisfied nor satisfied; 4) somewhat satisfied; 5) very satisfied.
Time Frame: 12 weeks post final treatment
Population: All subjects completing the satisfaction questionnaire are included in the analysis population. Subject responses deemed inconclusive or not answered were excluded from the satisfactions counts.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 15
Participants
  Procedure comfortable to very comfortable | 13
  Somewhat to very visible fat reduction | 6
  Overall treatment effect about or more than expect | 5
  Would recommend to a friend | 4

4. Secondary Outcome: Change in the Fat Layer Thickness
Description: Caliper measurements will be obtained prior to treatment and at the 12-week follow-up visit to assess for changes to the fat layers in the flanks. After the treatment area is identified and marked, the thickness of fat layer will be measured using a caliper at the middle of the fat bulge. For each treatment area, three (3) measurements will be taken and recorded. The average of the three measurements will be calculated. The location of where measurements were taken will be recorded on a transparency sheet along with reference points using the subject's body landmarks (such as a mole, skin pigmentation). This transparency will be used at post treatment visit to locate the measurement sites. Results will be reported in millimeters of fat layer.
Time Frame: Pre-treatment and 12 weeks post-final treatment
Population: Subjects included in the analysis population received CoolSculpting on both flanks and that had evaluable caliper measurements obtained pre-treatment and at 12 week post treatment.
Measure: Mean (Standard Deviation); unit: millimeters of fat
Units Other Than Participants: Treatment areas
Arm/Group | CoolSculpting Treatment Group
Number analyzed (Participants) | 15
Number analyzed (Treatment areas) | 29
millimeters of fat | -1.4 (1.7)

5. Secondary Outcome: Operator Feedback
Description: Operator performing or assisting with study procedure will complete two questionnaire at the treatment visit regarding the fit of two applicators: 1) CoolCurve+ and 2) CoolCurve The questionnaire consists of four multiple choice questions, each having a 5-point scale, with '5' representing the best and '1' the worst.
Time Frame: Pre-treatment/treatment day
Population: The operators using the device and applicators in the study participated in, or provided treatment using the Cool Curve and the CoolCurve+ applicator.
Measure: Number; unit: score on a scale
Groups:
- Operator Feedback on CoolCurve Applicator; Operator Feedback on CoolCurve + Applicator: The operator assessed the fit and tissue draw into each of 2 applicators. The assessment was done using a multiple choice questionnaire for each applicator type.
Arm/Group | Operator Feedback on CoolCurve Applicator | Operator Feedback on CoolCurve + Applicator
Number analyzed (Participants) | 15 | 15
score on a scale | 3.20 | 4.47

ADVERSE EVENTS:
Time Frame: Adverse event reports are solicited from the time of enrollment through the 12 week follow-up visit.
Description: Adverse events (AE) will be assessed continuously throughout the study. An adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device.
Arm/Group | CoolSculpting Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No